CLINICAL TRIAL: NCT00494676
Title: Community-based Multi-center Randomized Control Trial of Peripheral Prism Glasses for Hemianopia
Brief Title: Clinical Trial of Peripheral Prism Glasses for Hemianopia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Alexandra Bowers (Other)
Collaborators: Chadwick Optical Inc. (Industry); National Eye Institute (NEI) (NIH)
Responsible Party: Sponsor-Investigator, Alexandra Bowers, Principal Investigator, Schepens Eye Research Institute
Organization: Massachusetts Eye and Ear Infirmary (Other)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 2006-016; R44EY014723 (NIH)
Record Dates: First submitted 2007-06-28; First posted 2007-07-02 (Estimated); Results first posted 2013-09-13 (Estimated); Last update posted 2017-04-04 (Actual); Status verified 2017-04

CONDITIONS: Homonymous Hemianopia
Keywords: Hemianopia; Mobility; Rehabilitation; Low vision
MeSH Terms: conditions — Hemianopsia; Vision, Low

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Real prism glasses first, then sham (Experimental): Participants in this arm will receive high power (57 prism diopter) peripheral prism glasses in the first period of the crossover and low power sham peripheral prism glasses in the second period
  Interventions: Device: High power (57 prism diopter) peripheral prism glasses; Device: Low power sham peripheral prism glasses
- Sham prism glasses first, then real (Experimental): Participants in this arm will receive low power sham peripheral prism glasses in the first period of the crossover and high power (57 prism diopter) peripheral prism glasses in the second period
  Interventions: Device: High power (57 prism diopter) peripheral prism glasses; Device: Low power sham peripheral prism glasses

INTERVENTIONS:
Device: High power (57 prism diopter) peripheral prism glasses — All patients will wear two pairs of prism glasses in a crossover design: the high power peripheral prism glasses and sham peripheral prism glasses. Each pair of prism glasses will be worn for four weeks
Device: Low power sham peripheral prism glasses — Low power (5 prism dioptre) prism glasses that provide only about 2 degrees of visual field expansion.

SUMMARY:
The purpose of this study is to evaluate the functional utility for general mobility (walking) of new high power permanent peripheral prism glasses, which provide visual field expansion device for patients with homonymous hemianopia (the complete loss of half the field of vision on the same side in both eyes). The efficacy of real peripheral prism glasses will be assessed relative to sham peripheral prism glasses.

DETAILED DESCRIPTION:
Patients with hemianopic field loss are unaware of objects in their blind (non-seeing) hemi-field and often experience difficulties with mobility and navigation, such as walking into obstacles on the side of the field loss. In 2000, Peli (2000) described a new peripheral-prism design of prismatic correction for hemianopia, which addresses many of the inadequacies of existing designs of hemianopic visual aids, and produces true field expansion (i.e. the simultaneously seen field is larger with the device than without). In collaboration with the Schepens Eye Research Institute (Boston, MA), Chadwick Optical Inc (White River Junction, VT) has developed a permanent form of Fresnel prism segments, which are made from an acrylic material and can be embedded in a plastic spectacle lens. These permanent prisms offer better cosmesis, optical quality and durability than the temporary 40 prism-diopter press-on Fresnel prism segments used in previous evaluations of the peripheral prism system.

In this study we will evaluate new high-power (57 prism diopter) permanent peripheral prism glasses. The study will employ a crossover design in which each participant will wear a pair of real prism glasses (high-power, 57 prism diopter) and a pair sham prism glasses (low-power, 5 prism diopters, that provide little field expansion) in counterbalanced order. The efficacy of the real prism glasses relative to the sham prism glasses will be assessed for general mobility (walking). We expect that participants will prefer the real prism glasses over the sham prism glasses as the former will be more helpful for obstacle detection when walking.

Prism glasses will be fitted by Low Vision Practitioners at community-based Vision Rehabilitation Clinics. After wearing the first pair of glasses for 4 weeks, participants will return for an in-office follow up visit, at which a questionnaire will be administered to record their experiences of wearing the glasses. The second pair of prism glasses will then be fitted. Another questionnaire will be administered 4 weeks later to record the experiences of wearing the second set of glasses.

At the end of the period of wearing the second pair of prism glasses, a clinical decision will be made as to whether the participant should continue to use the real prism glasses (e.g. if a participant finds the prism glasses helpful for obstacle avoidance when walking). For participants who continue with the prism glasses, a final telephone follow-up interview will be conducted after about 6 months.

ELIGIBILITY:
Inclusion Criteria:

* At least 18 years of age.
* Sighted in both eyes, with monocular visual acuity (best corrected vision), of at least 20/50 in each eye.
* Complete homonymous hemianopia of more than 3 months duration
* Refractive error within the -5 dioptre to +5 dioptre range
* No significant cognitive impairment
* No history of wearing the Peli system of peripheral prisms for hemianopic field expansion (patients who have worn another type of prismatic correction for hemianopia such as yoked prisms or the Gottlieb VAS system can participate in the study)
* No physical or mental disabilities, including cognitive dysfunction, balance problems or other deficits that could impair ability to walk or use the peripheral prism spectacles.
* Able to walk (using a cane or walker is OK) or control the movements of their own wheelchair.
* In sufficiently good health to attend four in-office visits.

Exclusion Criteria:

* Diagnosis of dementia
* Diagnosis of visual neglect
* History of seizures in the last 6 months
* Incomplete hemianopia

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 73 (Actual)
Dates: Start 2007-09; Primary Completion 2009-07 (Actual); Study Completion 2010-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Alex R Bowers, PhD, Principal Investigator — Schepens Eye Research Institute; Karen Keeney, MSBA, Principal Investigator — Chadwick Optical Inc.
Locations (13):
- United States (12):
  - UAB Center for Low Vision Rehabilitation, Birmingham, Alabama
  - Vista Center for the Blind and Visually Impaired, Palo Alto, California
  - Visual Health@Jupiter Eye Center, Jupiter, Florida
  - Emory Optical Low Vision, Atlanta, Georgia
  - Illinois Eye Institute, Chicago, Illinois
  - Indiana University School of Optometry, Low Vision Rehabilitation and Primary Care Services, Bloomington, Indiana
  - University of Kansas Medical Center, Prairie Village, Kansas
  - Schepens Eye Research Institute, Boston, Massachusetts
  - Vision Care Specialists, P.C., Southborough, Massachusetts
  - Academy Eye Associates, Durham, North Carolina
  - Seven Lakes Eye Care, West End, North Carolina
  - NSU Oklahoma College of Optometry,, Tahlequah, Oklahoma
- Manchester Royal Eye Hospital, Manchester, United Kingdom

REFERENCES:
- [Background] Peli E. Field expansion for homonymous hemianopia by optically induced peripheral exotropia. Optom Vis Sci. 2000 Sep;77(9):453-64. doi: 10.1097/00006324-200009000-00006. PMID 11014672
- [Background] Bowers AR, Keeney K, Peli E. Community-based trial of a peripheral prism visual field expansion device for hemianopia. Arch Ophthalmol. 2008 May;126(5):657-64. doi: 10.1001/archopht.126.5.657. PMID 18474776
- [Derived] Bowers AR, Keeney K, Peli E. Randomized crossover clinical trial of real and sham peripheral prism glasses for hemianopia. JAMA Ophthalmol. 2014 Feb;132(2):214-22. doi: 10.1001/jamaophthalmol.2013.5636. PMID 24201760
- See also: Dr Eli Peli's Vision Rehabilitation Lab at Schepens Eye Research Institute — http://www.eri.harvard.edu/faculty/peli/index.html

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited at 13 study sites, including Dr. Peli's lab at Schepens, 11 vision rehabilitation clinics in the US, and one in the UK. The clinics included university, hospital and private-practice clinics. Each site recruited a median of 7 participants (range 3 to 12). Data were collected in the period October 2007 to January 2010.
Pre-assignment Details: 97 subjects were screened for eligibility of which 73 met the study criteria and were enrolled. The main reasons for not meeting the inclusion criteria were incomplete hemianopia and spatial neglect.
Groups:
- Real Prism Glasses Then Sham: Real prism glasses for 4 weeks followed by sham prism glasses for 4 weeks
- Sham Prism Glasses Then Real: Sham prism glasses for 4 weeks followed by real prism glasses for 4 weeks
Period: Allocation
Arm/Group | Real Prism Glasses Then Sham | Sham Prism Glasses Then Real
Started | 37 | 36
Completed | 35 | 32
Not Completed | 2 | 4
Not completed — Withdrawal by Subject | 2 | 4
Period: First Intervention
Arm/Group | Real Prism Glasses Then Sham | Sham Prism Glasses Then Real
Started | 35 | 32
Completed | 34 | 29
Not Completed | 1 | 3
Not completed — Withdrawal by Subject | 1 | 3
Period: Second Intervention
Arm/Group | Real Prism Glasses Then Sham | Sham Prism Glasses Then Real
Started | 34 | 29
Completed | 33 | 28
Not Completed | 1 | 1
Not completed — Withdrawal by Subject | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Entire Study Population: Includes groups allocated to receive real prism glasses first and sham prism glasses first
Arm/Group | Entire Study Population
Number analyzed (Participants) | 73
Age, Continuous [Mean (Standard Deviation); unit: years] | 56 (16)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 26
  Male | 47
Duration of hemianopia [Median (Inter-Quartile Range); unit: Months] | 18 [8 to 38]
Side of hemianopia [Number; unit: Participants]
  Right hemianopia | 25
  Left hemianopia | 48

OUTCOME MEASURES:

1. Primary Outcome: Overall Proportion Saying "Yes" to Real Prism Glasses
Description: At the end of each crossover period, participants were asked a yes/no question: "If the study were to end today, would you want to continue with these prism glasses (i.e. the prism glasses worn in that period)?" The primary outcome was the overall difference, across the two periods of the crossover, between the proportion of participants saying "yes" to real prism glasses and the proportion saying "yes" to sham prism glasses.
Time Frame: Evaluated after 4 weeks of wearing each type of prism glasses
Population: Only participants who completed the crossover were included in this analysis
Measure: Number; unit: participants
Arm/Group | Entire Study Population
Number analyzed (Participants) | 61
participants
  Said yes to real prism glasses | 39
  Said yes to sham prism glasses | 22
Statistical Analysis 1: Comparison: Entire Study Population; The analysis used a McNemar test for data combined across both periods of the crossover. We estimated that 70% and 35% of participants would say yes to the real and sham prisms, respectively. For a 2-tailed test, the minimum sample size to detect a 35% difference in yes responses to real and sham prisms was 57 participants, assuming 30% overlap (30% said yes to both pairs of glasses), power of 90% and α of 1%. Assuming an attrition rate of 20%, we planned to enroll 68 participants; Test type: Superiority or Other; p = 0.001, McNemar; Odds Ratio (OR) = 5.2, 95% CI 2-sided [1.8 to 21.0] — The marginal odds ratio based on discordant pairs was computed

2. Secondary Outcome: Mobility Change Score (All Participants Who Completed Crossover)
Description: Perceived difficulties with mobility were quantified using a 5-point rating scale (no difficulty to extreme difficulty) for 7 situations (items) relevant to people with hemianopia, including at home, in stores, outdoors, in unfamiliar areas, in familiar areas, in crowded areas, and noticing objects off to the side when walking. The questionnaire was administered at baseline (without prisms) and after each period of the crossover. Interval scale measures of perceived difficulty with overall mobility for each participant were estimated using Rasch analysis of the responses to all seven items (Winsteps software, version 3.70.0.226). Rasch measures were expressed as logits (log odds ratios). Mobility change scores for real and sham prisms were defined as the difference in perceived difficulty relative to baseline (in logits).
Time Frame: Evaluated after 4 weeks of wearing each type of prism glasses
Population: Only participants who completed the crossover were included in this analysis
Measure: Mean (Standard Deviation); unit: logits
Arm/Group | Entire Study Population
Number analyzed (Participants) | 61
logits
  Mobility change score for real prisms | 1.9 (3.3)
  Mobility change score for sham prisms | 1.3 (2.5)
Statistical Analysis 1: Comparison: Entire Study Population; Mobility improvement scores were normally distributed. A paired t-test was used to conduct a within-subjects comparison of the crossover differences in mobility scores between real and sham prism glasses. An alpha level of 5% was used to indicate statistical significance for secondary analyses; Test type: Superiority or Other; p = 0.09, t-test, 2 sided; Mean Difference (Final Values) = 0.6, 95% CI 2-sided [-0.1 to 1.3], Standard Deviation 2.6

3. Secondary Outcome: Mobility Change Score (Only Participants Who Continued Prism Wear in the Long Term)
Description: as for outcome 2
Time Frame: Evaluated after 4 weeks of wearing each type of prism glasses
Population: This is a subgroup analysis of the mobility change scores for real and sham prism glasses evaluated during the crossover. The subgroup includes only those participants who completed the crossover and continued to wear prism glasses in the long term.
Measure: Mean (Standard Deviation); unit: logits
Groups:
- Entire Study Population Who Continued: Includes groups allocated to receive real prism glasses first and sham prism glasses first
Arm/Group | Entire Study Population Who Continued
Number analyzed (Participants) | 25
logits
  Mobility change score for real prisms | 3.0 (3.2)
  Mobility change score for sham prisms | 1.1 (2.4)
Statistical Analysis 1: Comparison: Entire Study Population Who Continued; Test type: Superiority or Other; p = 0.002, t-test, 2 sided; Mean Difference (Final Values) = 1.9, 95% CI 2-sided [0.7 to 3.0], Standard Deviation 2.7

4. Secondary Outcome: Mobility Change Score (Only Participants Who Discontinued Prism Wear in the Long Term)
Description: Perceived difficulties with mobility were quantified using a 5-point rating scale (no difficulty to extreme difficulty) for 7 situations (items) relevant to people with hemianopia, including at home, in stores, outdoors, in unfamiliar areas, in familiar areas, in crowded areas, and noticing objects off to the side when walking. The questionnaire was administered at baseline (without prisms) and after each period of the crossover. Interval scale measures of perceived difficulty with overall mobility for each participant were estimated using Rasch analysis of the responses to all seven items (Winsteps software, version 3.70.0.226). Rasch measures were expressed as logits (log odds ratios). Mobility improvement scores for real and sham prisms were defined as the difference in perceived difficulty relative to baseline (in logits).
Time Frame: Evaluated after 4 weeks of wearing each type of prism glasses
Population: This is a subgroup analysis of the mobility change scores for real and sham prism glasses evaluated during the crossover. The subgroup includes only those participants who completed the crossover and then discontinued wearing prism glasses.
Measure: Mean (Standard Deviation); unit: logits
Groups:
- Entire Study Population Who Discontinued: Includes groups allocated to receive real prism glasses first and sham prism glasses first
Arm/Group | Entire Study Population Who Discontinued
Number analyzed (Participants) | 35
logits
  Mobility change score for real prisms | 1.1 (3.3)
  Mobility change score for sham prisms | 1.6 (2.7)
Statistical Analysis 1: Comparison: Entire Study Population Who Discontinued; Test type: Superiority or Other; p = 0.21, t-test, 2 sided; Mean Difference (Final Values) = -0.5, 95% CI 2-sided [-1.2 to 0.3], Standard Deviation 2.1

ADVERSE EVENTS:
Arm/Group | Entire Study Population
Serious Adverse Events (participants affected / at risk) | 0/67
Other Adverse Events (participants affected / at risk) | 0/67

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes